CLINICAL TRIAL: NCT01352871
Title: The Effects of Concentration/Meditation on the Innate Immune Response During
Brief Title: The Effects of Concentration/Meditation on the Innate Immune Response During Human Endotoxemia
Status: Completed | Type: Observational
Sponsor: Radboud University Medical Center (Other)
Responsible Party: Professor P. Pickkers, Principle Investigator, Radboud University Nijmegen Medical Centre
Other Study IDs: LPS-concentration
Record Dates: First submitted 2010-11-26; First posted 2011-05-12 (Estimated); Last update posted 2011-06-07 (Estimated); Status verified 2011-02

CONDITIONS: Innate Immune Response
Keywords: Immunity, Innate; Attention; Concentration
MeSH Terms: interventions — Meditation; Lipopolysaccharides; Endotoxins

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (1):
- Concentration / meditation: The subject will try to influence the innate immune response by concentration / meditation in advance of and during endotoxemia
  Interventions: Behavioral: Concentration / meditation; Drug: lipopolysaccharide

INTERVENTIONS:
Behavioral: Concentration / meditation — from 30 minutes before endotoxin administration to 1,5 hrs after endotoxin administration the subject is concentrating / meditating with the goal to influence the innate immune response
Drug: lipopolysaccharide — lipopolysaccharide 2ng/kg intravenously
  Other Names: LPS; endotoxin

SUMMARY:
The innate immune response is the first line of defense against invading pathogens. Ideally, the inflammatory response is tightly regulated leading to both adequate protection to invading pathogens as well as limitation of an exuberant or unwanted immune response such as seen in sepsis or auto-immune diseases. It has become increasingly clear that the autonomic nervous system (ANS) and the innate immune response are intimately linked. Activation of the sympathetic division of ANS dampens inflammation via β2-adrenoceptors. On the other hand, in some cases, sympathetic drive can also stimulate the inflammatory response via α2-adrenoceptors. The parasympathetic branch of the ANS modulates the inflammatory response as well, since it was discovered that electrical stimulation of the efferent vagus nerve in rats greatly inhibits the innate immune response. Generally, the ANS is regarded as pure autonomic which can not be influenced by behavior. However, trough special concentration/mediation techniques mastered by certain individuals, it might be possible to modulate ANS activity. In addition, recent unpublished findings indicate that these concentration/meditation techniques can also influence the inflammatory response ex vivo.

In this study the investigators wish to investigate the effect of concentration/meditation on the innate immune response in vivo. In addition the investigators wish to elucidate the mechanism via which this effect is mediated. The investigators aim to use the so called human endotoxemia model. This model permits elucidation of key players in the immune response to a gram negative stimulus in vivo, therefore serving as a useful tool to investigate potential novel therapeutic strategies in a standardized setting.

Objectives:

Primary objective: The primary objective of the study is to determine the effect of concentration/meditation on the innate immune response induced by a lipopolysaccharide (LPS) challenge.

Secondary Objective(s):

1. To determine the effects of concentration/meditation on ANS activity. Electroencephalography (EEG), heart-rate variability (HRV), muscle sympathetic nerve activity and plasma concentrations of catecholamines will be measured for this purpose.
2. To determine if concentration/meditation can attenuate (subclinical) renal damage known to occur during human endotoxemia, markers of proximal and distal tubular damage will be measured at various time points.

ELIGIBILITY:
Inclusion Criteria:

* 45 - 55 years of age
* male
* Healthy

Exclusion Criteria:

* Use of any medication.
* Smoking.
* Bleeding disorder.
* Previous spontaneous vagal collapse.
* History, signs or symptoms of cardiovascular disease.
* Cardiac conduction abnormalities on the ECG consisting of a 2nd degree atrioventricular block or a complex bundle branch block.
* Hypertension (defined as RR systolic > 160 or RR diastolic > 90).
* Hypotension (defined as RR systolic < 100 or RR diastolic < 50).
* Renal impairment (defined as plasma creatinin >120 μmol/l).
* Liver enzyme abnormalities or positive hepatitis serology.
* Positive HIV serology or any other obvious disease associated with immune deficiency.
* Febrile illness in the week before the LPS challenge.
* Participation in another drug trial or donation of blood 3 months prior to the planned LPS challenge.

Ages: 45 Years to 55 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: One healthy male volunteer that masters the concentration/meditation technique.
Sampling Method: Non-Probability Sample
Enrollment: 1 (Estimated)
Dates: Start 2011-03; Primary Completion 2011-04 (Actual); Study Completion 2011-05 (Actual)

PRIMARY OUTCOMES:
Change in Plasma TNF-alpha levels | 0; 1; 1.5; 2; 3; 4; 6; 8; 12; 24 hrs after endotoxin administration
  Concentration of circulating TNF-alfa at certain timepoints.

SECONDARY OUTCOMES:
Change in plasma IL-6, IL-10 and IL-1ra levels and leukocyte counts | 0; 1; 1.5; 2; 3; 4; 6; 8; 12; 24 hrs after endotoxin administration
  circulating IL-6, IL-10 and IL-1ra levels at certain timepoints.
  Leucocyte count and differentiation will be measured
Change in measures of autonomous nervous system activity | at regulare intervals before and during endotoxemia
  * Electroencephalography (EEG)
  * Heart rate variability (HRV)
  * Plasma cathecholamines
  * Muscle sympathetic nerve activity (MSNA)
Change in markers of subclinical renal tubular damage | before and at 0-3, 3-6, 6-9, 9-12 and 12-24 hrs after endotoxemia
  determination of markers in urine collected within the above mentioned intervals.
  GSTA1-1 will be used as marker for proximal tubular damage GSTP1-1 will be used as marker for distal tubular damage

CONTACTS AND LOCATIONS:
Overall Officials: Peter Pickkers, MD, PhD, Principal Investigator — Radboud University Medical Center
Locations (1):
- Radboud University Nijmegen Medical Centre, Nijmegen, Gelderland, Netherlands